CLINICAL TRIAL: NCT06925594
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Human TH-SC01 Cell Injection in the Treatment of Anal Fistulas in Patients With Non-active/Mildly Active Crohn's Disease
Brief Title: Phase 3 Study of Human TH-SC01 Cell Injection for Treating Perianal Fistulas in Patients With Crohn's Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TH-SC01-CD-Ⅲ-01
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): 120 million cells administered by intralesional injection.
  Interventions: Other: Human TH-SC01 cell injection
- Placebo-control group (Placebo Comparator): 24 mL saline solution by intralesional injection
  Interventions: Other: Saline solution

INTERVENTIONS:
Other: Human TH-SC01 cell injection — Human TH-SC01 cell injection is a cell suspension in aseptic buffered solution containing human expanded umbilical cord-derived stem cells of allogeneic origin in disposable vials with no preservative agents. The cells will be given at a dose of 120 million cells (5 million cells / mL) for intralesional injection.
  Arms: Treatment Arm
Other: Saline solution — Placebo (saline solution) will be given also for intralesional injection at the same quantity (volume, 24 mL) and following the same schedule.
  Arms: Placebo-control group

SUMMARY:
The purpose of this study is to evaluate the efficacy of human TH-SC01 cell injection for the treatment of perianal fistulas in Crohn's Disease over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Subjects with Crohn's disease diagnosed at least 6 months earlier according to the Chinese Consensus Opinion on the Diagnosis and Treatment of Inflammatory Bowel Diseases (Beijing, 2018)
3. Subjects with active perianal fistula and non active luminal CD defined by a CDAI ≤ 200.
4. Presence of perianal fistulas with a maximum of 2 fistulas (internal openings) and a maximum of 3 external openings, assessed by clinical assessment and MRI.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
6. American Society of Anesthesiologists (ASA) physical status classification of grade I to grade II.
7. All subjects and their partners were not planning to have a child from screening to the end of the trial and agreed to use effective non-drug contraception during the trial.

Exclusion Criteria:

1. Subjects allergic to human serum albumin, human platelet lysate, gentamicin sulfate, anesthetic drugs or MRI contrast agents.
2. Subjects with active infection evaluated by the investigator
3. Subjects with active Crohn's disease before drug administration or have not completed the induction-phase treatment.
4. Subjects with abscess or collections >2 cm.
5. Rectal and/or anal stenosis , if this means a limitation for any surgical procedure
6. Subjects with concurrent active proctitis.
7. Subjects with other fistulas such as rectum/anal canal-vaginal fistulas or rectum-bladder fistulas.
8. Patients have undergone a diverting stoma operation in the past, except for patients have completed stoma closure at least one month before drug administration.
9. Patients plan to undergo surgery in the perianal area during the trial period due to other diseases other than anal fistula.
10. Subjects with abnormal laboratory results: liver function: total bilirubin >=1.5 × ULN, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >=2 × ULN; renal function: creatinine clearance below 60 mL/minute calculated using Cockcroft-Gault formula or by serum creatinine >=1.5 × upper limit of normal (ULN).
11. Serum virology test (HBeAg, HCV antibody, HIV antibody, Treponema pallidum antibody) positive.
12. Subjects with malignant tumors or a history of malignant tumors.
13. Subjects with congenital or acquired immunodeficiency.
14. Contraindication to MRI scan
15. Current or recent history of abnormal, severe, progressive, uncontrolled hepatic, haematological, gastrointestinal (except CD), endocrine, pulmonary, cardiac, neurological, psychiatric, or cerebral disease.
16. Subjects received stem cell treatment within two years prior to screening.
17. Patient with ongoing steroid treatment or treated with steroids in the last 4 weeks.
18. Patient undergone major surgical operations (such as orthopedic surgery, abdominal surgery) within one month before drug administration, or Patient plan to receive surgeries during the study period (except for the surgeries required by the procedures of this trial).
19. Patients with a history of drug abuse or alcoholism (Criteria for alcoholism: having a long-term drinking history of more than 5 years, with the amount of ethanol equivalent to ≥40g/d for men and ≥20g/d for women, or having a history of heavy drinking within 2 weeks, with the amount of ethanol equivalent to >80g/d. The conversion formula for the amount of ethanol (g) = the amount of alcohol consumed (ml) × the ethanol content (%) × 0.8).
20. Pregnant or lactating women.
21. Patients with a history of diverting ostomy, except those who have undergone stoma reversal at least 1 month prior to drug administration.
22. Other diseases or conditions that the investigator deems inappropriate for participating in this clinical trial, such as poor subject compliance and the expectation of being unable to complete follow-up and evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2028-06-28 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects achieved combined remission | 24 weeks
  Combined Remission of perianal fistulising Crohn's disease defined as the all treated external openings achieved clinical remission at week 24， and absence of collections > 2 cm of the treated perianal fistulas confirmed by centrally blinded MRI assessment by week 24.

SECONDARY OUTCOMES:
The proportion of subjects achieved clinical remission | 24 weeks ，52 weeks and104 weeks
  Clinical Remission defined as closure of all treated external openings that were draining at baseline despite gentle finger compression, and no obvious fistulas can be felt by digital examination，as clinically assessed.
The proportion of subjects achieved a clinical response | 24 weeks，52 weeks and104 weeks
  Clinical response defined as closure of at least 50% of all treated external openings that were draining at baseline, as clinically assessed
The proportion of subjects recurrence | 24 weeks，52 weeks and104 weeks
  Recurrence defined as the reopening of the closed external openings that had achieved clinical remission after treatment, the appearance of spontaneous fluid drainage, or the presence of fistulas with fluid collections > 2 cm as assessed by enhanced pelvic MRI
Time to achieve clinical remission, clinical response and recurrence | 24 weeks，52 weeks and104 weeks
  Time to achieve clinical remission, clinical response and recurrence within 24 weeks after drug administration.
The proportion of subjects achieved combined remission | 52 weeks and104 weeks
  Combined Remission of perianal fistulising Crohn's disease at week 52 and 104 (as defined for week 24)
VAS score | 24 weeks，52 weeks and104 weeks
  Change from baseline in pain score (VAS score).Total score ranges from 0 to 10. Higher score means more pain
Perianal Disease Activity Index (PDAI) | 24 weeks，52 weeks and104 weeks
  Change from baseline in Perianal Disease Activity Index (PDAI). Total score ranges from 0 to 20. Higher score means more severe disease
Crohn's Disease Activity Index (CDAI) score | 24 weeks，52 weeks and104 weeks
  Change from baseline in the Crohn's Disease Activity Index (CDAI) score. Higher score means more severe disease and especially severe disease was defined as a value of greater than 450
Inflammatory Bowel Disease Questionnaire（IBDQ）score | 24 weeks，52 weeks and104 weeks
  Change from baseline in IBDQ score. Total score ranges from 32 to 224. Higher score means better quality of life
Anal sphincter function：Wexner incontinence score | 24 weeks，52 weeks and104 weeks
  Change from baseline in anal sphincter function, Wexner incontinence score,Total score ranges from 0 to 20. Higher score means more severe disease
peripheral blood cytokines | 2 weeks，4 weeks ，8 weeks ，12weeks and 24 weeks
  Changes in the levels of peripheral blood cytokines compared to the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Topcel-KH Pharmaceutical Co., Ltd., Nanjing, Jiangsu, China